CLINICAL TRIAL: NCT05728528
Title: Impact of Moderate to Vigorous-intensity Physical Activities on Pharmacokinetic-guided Extended Half-life FVIII Concentrates Prophylaxis Severe Hemophilia A Patients
Brief Title: Impact of Moderate Intensity Physical Activities on PK-guided EHL FVIII Concentrates Prophylaxis Severe HA Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Darintr Sosothikul, Associate Professor, Head of Integrative and Innovative Hematology/Oncology Research Unit at Faculty of Medicine, Chulalongkorn University., Chulalongkorn University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 996/2565
Record Dates: First submitted 2022-12-28; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PK-guided EHL FVIII concentrates prophylaxis with moderate intensity physical activities (Experimental): PK-guided EHL FVIII concentrates prophylaxis with moderate intensity physical activities
  Interventions: Drug: combination between moderate to vigorous-intensity physical activities and pharmacokinetic-guided extended half-life FVIII concentrates prophylaxis
- PK-guided EHL FVIII concentrates prophylaxis alone (Active Comparator): PK-guided EHL FVIII concentrates prophylaxis alone
  Interventions: Drug: pharmacokinetic-guided extended half-life FVIII concentrates prophylaxis alone

INTERVENTIONS:
Drug: combination between moderate to vigorous-intensity physical activities and pharmacokinetic-guided extended half-life FVIII concentrates prophylaxis — combination between moderate to vigorous-intensity physical activities and pharmacokinetic-guided extended half-life FVIII concentrates prophylaxis
  Arms: PK-guided EHL FVIII concentrates prophylaxis with moderate intensity physical activities
Drug: pharmacokinetic-guided extended half-life FVIII concentrates prophylaxis alone — pharmacokinetic-guided extended half-life FVIII concentrates prophylaxis alone
  Arms: PK-guided EHL FVIII concentrates prophylaxis alone

SUMMARY:
To compare clinical outcomes before and after using combination between moderate to vigorous-intensity physical activities and pharmacokinetic-guided extended half-life FVIII concentrates prophylaxis in moderate to severe hemophilia A patients

DETAILED DESCRIPTION:
This is a prospective cohort study of severe hemophilia A patients receiving low-dose EHL FVIII concentrates with PK-guided EHL FVIII concentrates prophylaxis alone for 6 months. Additional exercise workshops from sport scientists were introduced individually to this group of patients along with using the same prophylaxis method for another period of 6 months. The annualized bleeding rates (ABR), the annualized joint bleeding rates (AJBR), the haemophilia-specific quality-of-life (Haemo-QoL-A) scores, the hemophilia Joint Health Scores (HJHS) and skeletal muscle mass were compared between these two periods

ELIGIBILITY:
Inclusion Criteria:

* Severe Hemophilia A patients

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
annualized bleeding rates (ABR) | 6 months
  annualized bleeding rates (ABR)
annualized joint bleeding rates (AJBR) | 6 months
  annualized joint bleeding rates (AJBR)
haemophilia-specific quality-of-life (Haemo-QoL-A) scores | 6 months
  haemophilia-specific quality-of-life (Haemo-QoL-A) scores
hemophilia Joint Health Scores (HJHS) | 6 months
  hemophilia Joint Health Scores (HJHS)

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srichumpuang C, Rakmanotham A, Moonla C, Sosothikul D. Moderate- to vigorous-intensity physical activities for hemophilia A patients during low-dose pharmacokinetic-guided extended half-life factor VIII prophylaxis. Orphanet J Rare Dis. 2024 Mar 26;19(1):135. doi: 10.1186/s13023-024-03092-2. PMID 38532451